CLINICAL TRIAL: NCT02080832
Title: Brain Function and Structure in Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM15378; 2P50DA009262-16A1 (NIH)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Cocaine Dependence
Keywords: substance abuse; cocaine; impulsivity; serotonin; MRI
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Impulsive Behavior | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Medication (Citalopram 20mg) (Experimental): Citalopram (20mg dose)
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Medication (Citalopram 40mg) (Experimental): Citalopram 40mg dose
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Citalopram — 20 mg or 40 mg daily for 8 weeks
  Other Names: Celexa; Citalopram HBr
  Arms: Medication (Citalopram 20mg); Medication (Citalopram 40mg)
Drug: Placebo — Placebo daily for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the role of brain MRI findings in predicting treatment outcomes among individuals with cocaine dependence.

DETAILED DESCRIPTION:
The Specific Aims of this project are:

Aim 1: To determine whether pretreatment brain activation on fMRI while performing a Go-Nogo task predicts response to pharmacotherapy in cocaine dependent subjects.

Hypothesis related to Aim 1:

Pretreatment fMRI BOLD activation in cocaine dependent subjects during impulsive responding on the Go-Nogo task predicts 8-week outcome from medication known to enhance serotonin function (citalopram). The regression coefficient of TES on pretreatment mean BOLD activation on the Go-Nogo task will be significantly greater for the citalopram group than the placebo group.

Aim 2: To determine whether pretreatment brain activation on fMRI while performing an attentional bias (cocaine Stroop) task predicts response to pharmacotherapy in cocaine dependent subjects.

Hypothesis related to Aim 2:

Pretreatment fMRI BOLD activation in cocaine dependent subjects during cocaine related words on the cocaine Stroop task predicts 8-week outcome from medication known to enhance serotonin function (citalopram). The regression coefficient of TES on pretreatment mean BOLD activation from the cocaine Stroop task will be significantly greater for the citalopram group than the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 18 to 50 who meet current DSM-IV criteria for cocaine dependence who are seeking treatment.

Exclusion Criteria:

1. Current DSM-IV diagnosis of any psychoactive substance dependence other than cocaine, marijuana, nicotine, or alcohol
2. Have a DSM-IV axis I psychiatric disorder or neurological disease or disorder requiring ongoing treatment and/or making study participation unsafe
3. Significant current suicidal or homicidal ideation
4. Medical conditions contraindicating citalopram pharmacotherapy (liver disease, seizure disorder, bleeding disorder, or prolonged QT interval on EKG)
5. Taking CNS active concomitant medications
6. Taking medications known to have significant drug interactions with the study medication
7. Having conditions of probation or parole requiring reports of drug use to officers of the court
8. Impending incarceration
9. Pregnant or breast feeding for female patients
10. Inability to read, write, or speak English
11. Having plans to leave the immediate geographical area within 3 months
12. Unwillingness or not competent to sign a written informed consent form
13. Individuals who have pacemakers, metal or electromechanical implants or metallic foreign bodies
14. Patients who are known to be HIV positive will not be included due to possible CNS effects of HIV.
15. Alcohol withdrawal symptoms or history of significant previous alcohol withdrawal symptoms.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Moeller, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For some consented participants, the imaging scan (MRI) quality was not sufficient to include those participants in the outcome analysis. These participants are captured by the"excluded from analysis by MRI" category. fMRI data was only analyzed from participants who underwent MRI scans at UT Houston which can't be combined with MRI scans at VCU.
Groups:
- Medication Citalopram (20mg Dose): Citalopram (20mg dose)
  Citalopram: 20 mg daily for 8 weeks
- Medication Citalopram (40mg Dose): Citalopram (40mg dose) 40mg daily for 8 weeks
Period: Overall Study
Arm/Group | Medication Citalopram (20mg Dose) | Placebo | Medication Citalopram (40mg Dose)
Started | 15 | 17 | 22
Completed | 6 | 5 | 6
Not Completed | 9 | 12 | 16
Not completed — Excluded from analysis by MRI | 9 | 10 | 14
Not completed — Lost to Follow-up | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Medication Citalopram 20mg: Citalopram (20mg dose)
  Citalopram: 20 mg daily for 8 weeks
- Medication Citalopram 40mg: Citalopram (40mg dose) 40mg daily for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Medication Citalopram 20mg | Placebo | Medication Citalopram 40mg | Total
Number analyzed (Participants) | 15 | 17 | 22 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 22 | 54
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 5 | 9
  Male | 14 | 14 | 17 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 12 | 13 | 18 | 43
  Caucasian | 1 | 3 | 2 | 6
  Hispanic | 2 | 1 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 22 | 54

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use/Treatment Effectiveness Score (TES)
Description: Number of benzoylecgonine negative urines divided by the total number of urines collected
Time Frame: 8 weeks of treatment
Measure: Number; unit: percentage of negative urines
Arm/Group | Medication (Citalopram 20mg) | Placebo | Medication (Citalopram 40mg)
Number analyzed (Participants) | 6 | 5 | 6
percentage of negative urines | 6.6 | 8.3 | 29

2. Other Pre Specified Outcome: fMRI Brain Activation in Right Inferior Frontal Gyrus
Description: Brain activation on fMRI while participants undergo a Go/Nogo task. Percent of significant cluster in Statistical Parametric Mapping (SPM) for contrast of Hard Nogo minus Easy Nogo correlation with treatment effectiveness score.
Time Frame: Baseline
Measure: Number; unit: Percent of significant voxels in cluster
Groups:
- Citalopram (20mg or 40mg): Participants treated with citalopram, either 20mg or 40mg
Arm/Group | Citalopram (20mg or 40mg) | Placebo
Number analyzed (Participants) | 13 | 4
Percent of significant voxels in cluster | 83 | 0

3. Other Pre Specified Outcome: fMRI Brain Activation in Right Precentral Gyrus
Description: as for outcome 2
Time Frame: Baseline
Measure: Number; unit: percent of significant voxels in cluster
Arm/Group | Citalopram (20mg or 40mg) | Placebo
Number analyzed (Participants) | 13 | 4
percent of significant voxels in cluster | 9 | 0

4. Other Pre Specified Outcome: fMRI Brain Activation in Right Orlandic Operculum
Description: as for outcome 2
Time Frame: Baseline
Measure: Number; unit: percent of significant voxels in cluster
Arm/Group | Citalopram (20mg or 40mg) | Placebo
Number analyzed (Participants) | 13 | 4
percent of significant voxels in cluster | 8 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Medication (Citalopram 20mg) | Placebo | Medication (Citalopram 40mg)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/6

LIMITATIONS AND CAVEATS:
Results should be viewed with caution due to small sample size. Data was only analyzed from participants who underwent MRI scans at UT Houston as data could not be combined with MRI scans at VCU.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes